CLINICAL TRIAL: NCT04507906
Title: Safety and Efficacy of Nivolumab Combined With Anlotinib in Advanced Non-small Cell Lung Cancer Patients Previously Treated With Checkpoint Inhibitor-A Single Center and Exploratory Study
Brief Title: Nivolumab Combined With Anlotinib as Re-challenge Treatment in Advanced NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Baohui Han, Director of pulmonary department of Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS2025
Record Dates: First submitted 2020-08-08; First posted 2020-08-11 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: NSCLC Stage IV; Checkpoint Inhibitor
Keywords: NSCLC; Nivolumab; Anlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab + Anlotinib Arm (Other)
  Interventions: Drug: Nivolumab Combined with Anlotinib

INTERVENTIONS:
Drug: Nivolumab Combined with Anlotinib — In combination dose finding phase, Phase 1b will begin with Dose Level 1; anlotinib 12 mg/day orally (from days 1 to 14 in a 21-day cycle) and nivolumab (360mg q3w, intravenously) will be administered to eligible subjects on a 21-day treatment cycle. Two dose de-escalation steps are included: Dose Level 2 (anlotinib 10 mg/day orally, from days 1 to 14 in a 21-day cycle) and nivolumab 360mg q3w, intravenously) and Dose Level 3 (anlotinib 8 mg/day orally, from days 1 to 14 in a 21-day cycle) and nivolumab 360mg q3w, intravenously).If RP2D was reached in Part A, eligible patients would be enrolled and receive nivolumab (360mg q3w, intravenously) plus anlotinib (RP2D, QD from day 1 to 14 of a 21-day cycle) .

SUMMARY:
This is a phase Ib/IIa, open-label, single center study, aiming to investigate safety and efficacy of nivolumab (administered intravenously) in combination with anlotinib (administered orally) in immunotherapy-treated advanced NSCLC. The study has been designed to allow an investigation of the optimal combination dose and schedule while ensuring the safety of patients with intensive safety monitoring. There are two main parts to this study; Part A, combination dose finding and Parts B, dose expansion. Part B will either be initiated if RP2D reached in Part A, or not initiated if RP2D was not reached in Part A.

Part A has been designed to identify the recommended dose of combination of nivolumab plus anlotinib for further clinical evaluation based upon assessment of the safety and tolerability data collected during the first 21 days (cycle 1, 21 days per cycle). The 21-day assessment period was selected as the major toxicities leading to cessation of dose de-escalation in such Phase I oncology studies (haematological, gastrointestinal, liver enzymes) are anticipated to present within this duration. "3+3"design was used in the dose finding cohort.

If RP2D was reached in Part A, eligible patients would be enrolled and receive nivolumab (360mg q3w, intravenously) plus anlotinib (RP2D, QD from day 1 to 14 of a 21-day cycle) till disease progression (PD) withdraw of consent, or unacceptable toxicity to further evaluate the safety, tolerability and efficacy in terms of ORR , DCR, DOR, PFS and OS. The tumor response will be evaluated according to RECIST Version 1.1 every 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. According to the 8th edition of the AJCC/UICC TNM staging system for NSCLC, patients with locally advanced (stage III B/III C), metastatic or recurrent (stage IV) NSCLC confirmed by histology or cytology who are unable to undergo surgery and radical concomitant radiochemotherapy and are confirmed to have at least one measurable lesion according to RECIST 1.1.
2. Without active brain metastasis
3. Previously treated with ICIs with progressive disease.
4. Age ≥18 years and ≤75 years;
5. ECOG PS score: 0 to 1
6. Palliative radiotherapy must be completed 7 days before the first dose of study drugs;
7. The main organs function is normal, that is, the following criteria met:

   1. Good hematopoietic function, defined as absolute neutrophil count ≥1.5×109 /L, platelet count≥100 ×109 /L, hemoglobin ≥90g/L [no blood transfusion or no erythropoietin (EPO) dependence within 7 days before enrollment]
   2. Biochemical test results should meet the following criteria: BIL < 1.25 times the upper limit of normal value (ULN); ALT and AST < 2.5 × ULN; in case of liver metastases, ALT and AST < 5 × ULN; Cr ≤1.5×ULN or creatinine clearance (CCr) ≥60ml/min; Coagulation function is good, INR and PT ≤1.5 times ULN; if the subject is receiving anticoagulant treatment, PT should be within the prescribed range of use of anticoagulant drugs;
8. Women of child-bearing age should agree to take contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study and within 6 months after the study; non-breast-feeding patients whose serum or urinary pregnancy test should be negative; male patients should agree to take contraceptive measures during the study and within 6 months after the study.
9. Patients are voluntarily enrolled into the study, sign the informed consent form and have good compliance.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded:

1. Subjects with active CNS metastases are excluded. Subjects are eligible if CNS metastases are adequately treated and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrollment. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).
2. Small cell lung cancer (including mixed small cell and non-small cell lung cancer) or central squamous cell carcinoma with cavity;
3. With obvious hemorrhage symptom
4. With driver mutation (EGFR/ALK/ROS1) or mutation status are unknown
5. Patients who have not received IO as frontline treatment;
6. Patients who have grade 3 AEs when treated with IO
7. Patients with many factors affecting oral medication, such as dysphagia, gastrointestinal resection, chronic diarrhea and intestinal obstruction;
8. Patients who are known to have active brain metastases, spinal cord compression, carcinomatous meningitis, or brain or leptomeningeal disease diagnosed by CT or MRI at the time of screening;
9. Patients with severe and / or uncontrolled diseases, such as: unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months before randomization, severe uncontrolled arrhythmias; uncontrolled blood pressure (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
10. Active or uncontrolled serious infection;
11. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
12. Not completely controlled eye inflammation or eye infection, or any condition that may lead to the above-mentioned ocular diseases
13. Poorly controlled diabetes (fasting blood glucose (FBG) > 10mmol/L);
14. Routine urine test result indicates that urine protein ≥++, and 24-hour urine protein quantitation is confirmed to be > 1.0 g;
15. Active tuberculosis;
16. Uncontrolled hypercalcemia (> 1.5 mmol/L calcium ion or calcium > 12 mg/dL or corrected serum calcium > ULN), or symptomatic hypercalcemia requiring continued diphosphate therapy;
17. Long-term unhealed wounds or fractures;
18. Patients who have a history of psychotropic drug abuse and cannot abstain from it or have mental disorders;
19. Patients who are known to have severe allergies (≥ grade 3) to active ingredients and any excipients of dacomitinib
20. Patients who have other malignant tumors (except radical cervical carcinoma in situ, non-melanoma skin cancer, etc.) at the same time; patients who are evaluated by the investigator to have concomitant diseases that seriously endanger the safety of the patients or affect the patients completing the study.
21. The subjects or their sexual partners cannot or refuse to take effective contraceptive measures during the clinical trial
22. Pregnant or breast-feeding women
23. Previously treated including treated with traditional Chinese medicine
24. Patients who are allergic to any of the agent or any ingredient
25. Patients in other situations who are evaluated by the investigator to be ineligible to be enrolled

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6-9 weeks
  Patients who were assessed as partial response or complete response

SECONDARY OUTCOMES:
Disease control rate (DCR) | 6-9 weeks
  Patients who were assessed as partial response, complete response or stable disease
Progression-free survival (PFS) | 5-7 months
  Time from enrollment to progression or death
Overall survival (OS) | 13-15 months
  Time from enrollment to death of any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang B, Liu H, Shi C, Gao Z, Zhong R, Gu A, Chu T, Wang H, Xiong L, Zhang W, Zhang X, Yan B, Teng J, Wang W, Bai H, Qiao R, Cheng L, Kuang Y, Zhao R, Zhong H, Han B. Safety and efficacy of multi-target TKI combined with nivolumab in check-point inhibitor-refractory patients with advanced NSCLC: a prospective, single-arm, two-stage study. BMC Cancer. 2024 Jun 11;24(1):715. doi: 10.1186/s12885-024-12479-0. PMID 38862908